CLINICAL TRIAL: NCT02105623
Title: EARly Prevention of aTHeroma Progression
Acronym: EARTH
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow enrollement, Low Follow-up rate
Sponsor: CHEOL WHAN LEE, M.D., Ph.D (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, CHEOL WHAN LEE, M.D., Ph.D, MD, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMCCV2013-09
Record Dates: First submitted 2014-04-03; First posted 2014-04-07 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Coronary Arteriosclerosis
Keywords: Coronary Arteriosclerosis; rosuvastatin
MeSH Terms: conditions — Coronary Artery Disease | interventions — Standard of Care; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Therapy (Active Comparator): Risk factor control Diet Exercise
  Interventions: Behavioral: Standard Therapy
- Rosuvastatin therapy (Experimental): Risk factor control Rosuvastatin
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Behavioral: Standard Therapy — Risk factor control Diet Exercise for 24months
  Arms: Standard Therapy
Drug: Rosuvastatin — Risk factor control rosuvastatin 5mg/day for 24months
  Arms: Rosuvastatin therapy

SUMMARY:
The purpose of this study is to compare standard therapy (risk factor control, life style modification) versus standard therapy plus low-dose rosuvastatin therapy (5mg/day) on progression of coronary atherosclerosis in statin naive individuals who have mild CAD (nonobstructive coronary atherosclerotic plaques) and normal LDL (low-density lipoprotein) cholesterol levels(<130mg/dl).

ELIGIBILITY:
Inclusion Criteria:

* Men or women at least 35 years of age
* Mild CAD (nonobstructive coronary atherosclerotic plaques, lumen narrowing <50%) and CAC score <300 in at least one segment of proximal or mid-portion of major epicardial coronary arteries
* LDL cholesterol <130mg/dl

Exclusion Criteria:

* History of stable angina, or acute coronary syndrome
* History of transient ischemic attack, or stroke
* Chronic kidney disease (eGFR< 60ml/min)
* Diabetes mellitus with microvascular complications or insulin therapy
* Hypertriglyceridemia (triglyceride >500mg/dl)
* Any statin therapy in the past 4 weeks
* Planned cardiac surgery or planned major non-cardiac surgery within 6 months.
* Chronic disease requiring treatment with oral, intravenous, or intra-articular corticosteroids (use of topical, inhaled, or nasal corticosteroids is permissible).
* A diagnosis of cancer (other than superficial squamous or basal cell skin cancer) in the past 3 years or current treatment for the active cancer.
* Any clinically significant abnormality identified at the screening visit, physical examination, laboratory tests, or electrocardiogram which, in the judgment of the Investigator, would preclude safe completion of the study.
* Hepatic disease or biliary tract obstruction, or significant hepatic enzyme elevation (ALT or AST > 3 times upper limit of normal).
* History of adult asthma manifested by bronchospasm in the past 6 months, or currently taking regular anti-asthmatic medication(s).
* Unwillingness or inability to comply with the procedures described in this protocol.
* Positive pregnancy test (all female subjects of childbearing potential must have a urine ß-human chorionic gonadotropin(hCG) pregnancy test performed at Screening and/ or within 7 days prior to randomization) or is known to be pregnant or lactating.
* Hypersensitivity to Crestor
* Skeletal muscle disease
* Combination use with cyclosporine
* Galactose intolerance, Lapp lactose deficiency or glucose-galactose malabsorption
* Combination use of protease inhibitor

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Percent change in total atheroma volume(TAV) | 2 years
  Percent change in total atheroma volume(TAV) at region of interest defined as(TAV at 24 months-TAV at baseline)/(TAV at baseline)x 100

SECONDARY OUTCOMES:
Change in PAV(Percent atheroma volume) at region of interest | 2years
  Change in PAV(Percent atheroma volume) at region of interest(PAV at 24months-PAV at baseline)
Change in overall TAV | 2years
  Sum of TAV in all coronary segments
Change in TAV at region of interest | 2years
  TAV at 24months-TAV at baseline
Change in overall CAC(coronary artery calcification) score | 2years
  overall CAC score at 24months-overall CAC score at baseline
Change in number of segment of any coronary atherosclerotic plaques | 2years
Percent change from baseline in lipid levels | 2years

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
This is not a publicly funded trial.